CLINICAL TRIAL: NCT00520715
Title: Epidemiology and Risk Factors Study of the Carriage of Fluoroquinolone Resistant Bacteria in the Commensal Flora of Patients Hospitalised in Medical Wards
Brief Title: Epidemiology of Fluoroquinolone Resistance in Human Commensal Flora in Patients Hospitalised in Medical Wards
Status: Completed | Type: Observational
Sponsor: Association Pour le Recherche en Infectiologie et en Médecine Interne (Other)
Collaborators: Pr Bruno Fantin (Other)
Responsible Party: Principal Investigator, Dr Victoire de Lastours, MD, Association Pour le Recherche en Infectiologie et en Médecine Interne
Other Study IDs: FQ/EPI
Record Dates: First submitted 2007-07-11; First posted 2007-08-24 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Colonization; Multi Drug Resistant Bacteria; Hospitalized Patients
Keywords: fluoroquinolone resistance; commensal flora; carriage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients at hospital admission: Patients at hospital admission in medical wards on our tertiray care hospital (Hôpital Beaujon, Clichy, France).

SUMMARY:
Emergence of bacterial resistance to antibiotics, which is a major public health issue, appears to involve predominantly commensal flora. No data exists concerning risk factors for the carriage of fluoroquinolone resistant bacteria in the flora of hospitalised patients. We will conduct a prospective open study including all unselected patients hospitalised in medical wards of one hospital. Nasal, pharyngeal and rectal swabs will be performed upon admission as well as a review of potential risk factors, after patient's information and acceptance. Resistance testing aiming 3 pathogens (Staphylococcus, Streptococcus and E. coli) will be performed on all specimens, and a case control study will compare risk factors from the resistant and non-resistant groups, for each pathogen. A thousand patients should be included in a year's time. This work could help understand risk factors involved in the carriage of fluoroquinolone resistant pathogens, potentially responsible for invasive infections and inter-patient transmission of resistance. Limiting bacterial resistance and transmission is a goal that can be successfully undertaken only if resistance mechanisms, but also risk factors of acquiring resistant bacteria are better understood.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients admitted to the internal medicine, oncology, cardiology and geriatric unit of Beaujon Hospital, Clichy, France.
* patient agreement

Exclusion Criteria:

* Age < 18
* patient refusal or incapable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults patients at hospital admission hospital stay >24 hours informed consent required
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoire de Lastours, MD, Principal Investigator
Locations (1):
- Hôpital Beaujon, Clichy, Île-de-France Region, France

REFERENCES:
- [Derived] de Lastours V, Chau F, Tubach F, Pasquet B, Ruppe E, Fantin B. Independent behavior of commensal flora for carriage of fluoroquinolone-resistant bacteria in patients at admission. Antimicrob Agents Chemother. 2010 Dec;54(12):5193-200. doi: 10.1128/AAC.00823-10. Epub 2010 Sep 27. PMID 20876373